CLINICAL TRIAL: NCT07080008
Title: A Single Center, Open Label Pilot Study to Assess the Feasibility and Safety of Lumitrace Injection for Intraoperative Ureter Visualization Comparing White Light (WL) Fluorescence (BLUE) in Participants Undergoing Minimally Invasive Abdominopelvic Surgeries
Brief Title: Evaluation of Lumitrace for Visualizing Ureters During Abdominopelvic Surgeries
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 400-100
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Ureter Injury
Keywords: Relmapirazin; Lumitrace
MeSH Terms: interventions — relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 130 mg Lumitrace (Experimental): Participants will receive a single intravenous 130 mg dose of Lumitrace. Within 30 minutes of injection, the ureter visualization will be captured by the KARL STORZ POWER LED BLUE System using white light and fluorescence and the surgeon will rate ureter visualization for each illumination mode based on qualitative Likert Scales.
  Interventions: Drug: Lumitrace; Device: KARL STORZ POWER LED BLUE System

INTERVENTIONS:
Drug: Lumitrace — Administered as a bolus intravenous injection over 30 - 60 seconds
  Other Names: Relmapirazin; MB-102
Device: KARL STORZ POWER LED BLUE System — Imaging will be acquired within 30 minutes post Lumitrace administration. Following the initial endoscopic surgical incision, the surgeon will record the image assessments based on Likert Scales.

SUMMARY:
The goal of this clinical trial is to learn if Lumitrace and the KARL STORZ POWER LED BLUE System can be used for anatomic visualization of the ureters in participants undergoing laparoscopic abdominopelvic surgery.

The main questions it aims to answer are:

* To evaluate the feasibility and clinical utility of Lumitrace to provide ureter visualization when used in tandem with the KARL STORZ POWER LED BLUE System during laparoscopic abdominopelvic surgery
* To evaluate the safety and tolerability of a single intravenous dose of Lumitrace in participants undergoing laparoscopic abdominopelvic surgery

Participants will participate in a Screening visit that will take place within 28 days of the scheduled administration of Lumitrace.

Up to 10 participants will be enrolled and will receive a single intravenous 130 mg dose of Lumitrace. Within 30 minutes of injection, the ureter visualization will be captured by the KARL STORZ POWER LED BLUE System using white light and fluorescence and the surgeon will rate ureter visualization for each illumination mode based on qualitative Likert Scales.

A safety follow-up visit will occur within 14 ±7 days of Lumitrace administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years - male or female

   1. Eligible female non-pregnant subjects who are either not of child-bearing potential or willing to use adequate contraception during the trial
   2. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 30 days post-dose administration
   3. For women of child-bearing potential, the subject should have a negative serum pregnancy test on day of surgery, and agrees to one of the following acceptable contraceptive methods used consistently and correctly from the time of consent through 30 days after Lumitrace administration; i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system, or male partner sterilization
   4. Men will not donate sperm during the study and for 30 days following the last dose of Lumitrace
2. Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
3. Participant is scheduled to undergo minimally invasive laparoscopic abdominopelvic surgery that may require ureter(s) identification
4. eGFR≥60 mL/min/1.73m2

Exclusion Criteria:

1. Participant has any serious or uncontrolled physical or psychiatric condition that in the opinion of the investigator would limit the their ability to complete study requirements or may put the subject at increased risk, or compromise the interpretability of study results, which makes the participant unsuitable for study participation
2. Participant is anticipated to require ureteral stenting during surgery
3. Participant has an active urinary tract infection requiring antibiotic therapy
4. Participant has moderate to severe cardiac disease that limits daily functioning (New York Heart Association Class III to IV) or other medical conditions that would impact safety or study compliance
5. Participant has any clinically relevant laboratory abnormality that could contraindicate surgery in the opinion of the PI
6. Participant with body weight < 30 kilogram (kg)
7. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, Lumitrace or other related products (intolerance to a drug is not considered a drug allergy)
8. Participant has received any investigational therapy within 30 days or 5 half-lives, whichever is longer, prior to screening
9. eGFR <60 mL/min/1.73m2
10. Participants with positive serum pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Intra-participant difference in laparoscopic view of ureter conspicuity for white light (WL) versus fluorescence (BLUE) | Day of surgery
  Imaging will be acquired within 30 minutes post Lumitrace administration. Images from one or both ureters may be evaluated for anatomical visualization. Following the initial endoscopic surgical incision, the surgeon will record the image assessments based on the Likert Scales as follows.
  White light visibility will be measured using a 4-point scale where 0 represents not visible and 3 represents excellent visibility. For images collected using the BLUE setting, intensity will be graded based on the following: (0 = none; 1 = mild; 2 = moderate; and 3 = strong).

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon, Inc.
Locations (1):
- University of Missouri, Kansas, City, School of Medicine; Division of Urogynecology and Reconstructive Pelvic Surgery,, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No